CLINICAL TRIAL: NCT01840800
Title: Ultrasound Guided Nerve Block Combinations for Anterior Cruciate Ligament Reconstruction; Femoral, Saphenous and Obturator (Posterior Branch)Nerves.
Brief Title: USG Nerve Blocks for ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Borglum Neimann (Other)
Responsible Party: Sponsor-Investigator, Jens Borglum Neimann, Associate professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2-2012-063
Record Dates: First submitted 2013-02-19; First posted 2013-04-26 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; anterior cruciate ligament reconstruction; ultrasound guided nerve blocks; opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active FEM+ONP (Active Comparator): Nerveblock of n. femoralis (FEM) with 10 ml Ropivacaine 7.5 mg/ml and nerveblock of obturator nerveposterior branch (ONP) with 10 ml Ropivacaine 7.5 mg/ml.
  Interventions: Drug: Ropivacaine
- Active SAPH+ONP (Active Comparator): Nerveblock of n.saphenous (SAPH) with 5 ml Ropivacaine 7.5 mg/ml and nerveblock of obturator nerve, posterior branch (ONP) with 10 ml Ropivacaine 7.5 mg/ml
  Interventions: Drug: Ropivacaine
- Placebo (Placebo Comparator): Saline 9 mg/ml
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ropivacaine
  Arms: Active FEM+ONP; Active SAPH+ONP
Drug: placebo
  Arms: Placebo

SUMMARY:
Anterior cruciate ligament reconstruction is a routine surgical procedure. Traditional femoral/sciatic block combinations effectively reduce postoperative pain, but results in considerable motor blockade. The investigators aimed to evaluate postoperative pain relief and the degree of motor block with block combinations of femoral nerve (FEM) and obturator [posterior branch] nerve (ONP), versus saphenous nerve (SAPH) and ONP, versus placebo blocks with isotonic saline. All patients received standard patient controlled analgesia with morphine.Randomized, placebo-controlled and double-blinded clinical trial. Following IRB approval, 81 patients were planned to be randomized to one of three USG block combinations: Active FEM+ONP, active SAPH+ONP or no active blocks (sham blocks) Ropivacaine 0.75% was used for all active blocks following induction of general anaesthesia [propofol-remifentanil, laryngeal mask airway]. Primary outcome measure: Localized PACU pain scores (AUC) 0-6 hours postoperatively at rest.

Secondary outcome measures: Opioid consumption, opioid related side effects, PACU time, motor abilities of daily living scores [modified Barthel/100 index], perceived ill health [Short form-8] scores and degree of motor blockade [Jensen- Børglum motor test].

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Isolated primary ACL reconstruction in general anaesthesia with hamstring graft.
* ASA 1-3.
* Written and informed consent to study protocol.

Exclusion Criteria:

* ACL reconstruction with patellar tendon graft
* Uncooperative patients.
* Patients that do not understand or speak danish.
* Daily use of opioids equivalent to > 40 mg morphine.
* Allergic to Ropivacaine.
* Alcohol abusers
* Contraindications to general anaesthesia.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
NRS (pain score) | Area under the curve (AUC) 0-6 hours postoperatively
  Numerical rating scale(0-10)

SECONDARY OUTCOMES:
Opioid consumption | 0-6 hours postoperatively
  Opioid consumption (PCA pump - mg of morphine)
opioid related side effects | 0-6 hours postoperatively
  Nausea (0-3), vomiting (>10 ml)
PACU time | 0-6 hours postoperatively
  Minutes in PACU
Motor abilities of of daily living | 0-24 hours postoperatively
  Modified Barthel/100 index
Perceived ill health | 0-24 hours postoperatively
  Short-Form-8
Degree of motor block. | 0-6 hours postoperatively
  Jensen-Borglum motor test

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, department of anesthesiology, Copenhagen, Denmark